CLINICAL TRIAL: NCT06907823
Title: Comparison of Sevoflurane and Propofol on ANI in Patients Undergoing General Anesthesia: a Prospective Randomized Controlled Study
Brief Title: Comparison of Sevoflurane and Propofol on ANI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Jimin Lee, Clinical professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11-2025-003
Record Dates: First submitted 2025-03-28; First posted 2025-04-02 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Propofol; Sevoflurane; Analgesia Nociception Index
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane (Other)
  Interventions: Drug: Sevoflurane
- Propofol (Other)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — propofol anesthesia
  Arms: Propofol
Drug: Sevoflurane — sevoflurane anesthesia
  Arms: Sevoflurane

SUMMARY:
The goal of this clinical trial is to compare the effect of sevoflurane and propofol on analgesia nociception index(ANI) in patients undergoing general anesthesia. The main question it aims to answer is whether propofol anesthesia results in lesser ANI change to a nociceptive stimulation compared to sevoflurane.

DETAILED DESCRIPTION:
Patients will be allocated to either propofol or sevoflurane group. Nociceptive event will be defined as long-lasting tetanic stimulation, square-wave, duration of 30 seconds , amplitude of 50mA, frequency of 50 Hz. analgesia nociception index value and hemodynamic parameters will be recorded 1-minute before and after nociceptive event.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists physical status class I or II

Exclusion Criteria:

* history of drugs that can affect the central nervous system and autonomic nervous system, such as anticholinergics, betablockers, antidepressants..etc.
* history of allergic reaction to sevoflurane and/or propofol
* history of and/or family history of malignant hyperthermia
* neurodegenerative disorder
* psychiatric disorder
* arrhythmia
* diabetes mellitus
* drug abuse history

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
analgesia nociception index change | During anesthesia period
  analgesia nociception index value 1-minute before tetanic stimulation and 1-minute after tetanic stimulation

SECONDARY OUTCOMES:
Hemodynamic change | During anesthesia period
  Blood pressure change 1 minute before tetanic stimuation and 1 minute after tetanic stimulation
Hemodynamic change | During anesthesia period
  Heart rate change before 1-minute before nociceptive stimuli and 1-minute after nociceptive stimuli